CLINICAL TRIAL: NCT06960616
Title: Improving Clinical Efficiency by Reducing Scheduled Follow-ups Using Cochlear America's Population Mean Mapping Strategy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Principal Investigator, Julie G. Arenberg, CCC-A, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000034
Record Dates: First submitted 2025-03-11; First posted 2025-05-07 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Deafness; Cochlear Hearing Loss
MeSH Terms: conditions — Deafness; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Population mean mapping, without 1 week follow-up (Experimental): Reduction in the number of follow-up visits and new programming strategy.
  Interventions: Other: Changes in traditional follow-up; Other: Population mean mapping
- Population mean mapping, traditional follow-up (Experimental): New programming strategy
  Interventions: Other: Population mean mapping
- Traditional mapping*, without 1 week follow-up (Experimental): Reduction in the number of follow-up visits.
  Interventions: Other: Changes in traditional follow-up
- Traditional mapping, traditional follow-up (No Intervention): Traditional follow-up plan

INTERVENTIONS:
Other: Changes in traditional follow-up — Traditional follow-up includes the following visits after activation: 1-week, 1-month, 3-months, 6-months and 1 year. With the intervention used, the 1-week follow-up is removed.
  Arms: Population mean mapping, without 1 week follow-up; Traditional mapping*, without 1 week follow-up
Other: Population mean mapping — Traditional mapping at activation involves the measurement of at least 5 electrodes (both T-levels and C-levels). The intervention uses a population mean mapping strategy where there is a pre-set dynamic range of 46 CL with a spot check of C-levels.
  Arms: Population mean mapping, traditional follow-up; Population mean mapping, without 1 week follow-up

SUMMARY:
The study is about the importance of each follow-up visit after activating a new cochlear implant in addition to evaluating the effectiveness and efficiency of a new programming strategy from Cochlear Americas. Investigators are looking for patients who have recently selected Cochlear Americas as their cochlear implant manufacturer of choice for their upcoming surgery. The aim of this study is to determine if 1) patient outcomes remain stable when reducing follow-up appointments and 2) Cochlear's population mean mapping can produce similar outcomes with patients while additionally reducing appointment times. The hypothesis is that using population mean mapping and reducing the number of follow-up visits after activation will yield similar performance outcomes to a standard of care while decreasing the length of appointment times and number of appointments needed for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Postlingually deafened
* Adults (18+)
* New cochlear implant recipients with Cochlear Americas devices; identified prior to activation
* Able to perform follow-up testing tasks (repeating words/sentences, indicating they heard a sound stimulus, completing questionnaires)
* English speakers

Exclusion Criteria:

* Patients who select other cochlear implant manufactured devices
* Pre-lingually deafened
* Multiple disabilities
* Unable to perform follow-up testing tasks (repeating words/sentences, indicating they heard a sound stimulus, completing questionnaires)
* Non-English speakers
* Children under the age of 18

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Speech perception scores | 1-year
  Speech perception scores via CNC word lists (percentages) at each visit. Scores are from 0 to 100% with 100% being the best.
Duration of programming session | 1-year
  Time spent programming (seconds) at each visit

SECONDARY OUTCOMES:
Quality of Life questionnaire | 1-year
  Patient outcomes via the Cochlear Implant Quality of Life-35 Profile questionnaire at each visit. Scores are out of 35 points and higher scores indicate better quality of life.
Soundfield detection thresholds | 1-year
  Change in soundfield detection thresholds (dB HL) between each visit. Detection thresholds should be between 20 and 35 dB HL and anywhere in that range is good.
programming levels | 1-year
  Change in programming levels between each visit (converted measure from CL to charge units). There is no indication of good and bad with programming levels, we are just measuring what they are and how stable they are over time.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Arenberg, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Mass Eye and Ear, Boston, Massachusetts, United States